CLINICAL TRIAL: NCT02102113
Title: Probing the Cannabinoid System in Individuals With a Family History of Psychosis
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1310012948
Record Dates: First submitted 2014-03-26; First posted 2014-04-02 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2024-08

CONDITIONS: Psychosis; Cannabis Use; THC; Marijuana; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Marijuana Abuse; Schizophrenia | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Family History of Psychosis (FHN) (Other): Individuals recruited with no history of psychosis in the family. They will receive the placebo, very low dose THC, and low dose THC interventions.
  Interventions: Drug: Placebo; Drug: Very Low Dose THC; Drug: Low Dose THC
- Family History of Psychosis (FHP) (Experimental): Individuals with a family member with a confirmed diagnosis of psychosis. They will receive the placebo, very low dose THC, and low dose THC interventions.
  Interventions: Drug: Placebo; Drug: Very Low Dose THC; Drug: Low Dose THC

INTERVENTIONS:
Drug: Placebo — placebo
Drug: Very Low Dose THC — Subjects will receive 0.010mg/kg.
  Other Names: delta 9-tetrahydrocannabinol
Drug: Low Dose THC — Subjects will receive 0.018 mg/kg over 20 minutes.
  Other Names: delta 9-tetrahydrocannabinol

SUMMARY:
The overall purpose of this study is to determine whether a family history of psychosis is associated with an altered cannabinoid system. This will be tested by studying individuals with and without a family history of psychosis and comparing their responses to delta 9-tetrahydrocannabinol (THC), a probe of the cannabinoid system. We hypothesize, that compared to controls with no family history of psychoses, individuals with a family history of psychoses will have an altered response to THC.

ELIGIBILITY:
Inclusion Criteria FHP:

* Exposure to cannabis at least once in their lifetime
* Medically and psychiatrically healthy based on screening
* Having one relative with a confirmed psychotic disorder

Exclusion Criteria FHP:

* Current or lifetime major DSM-IV Axis I disorder
* Current or lifetime treatment (at least 6 months) with psychotropic medications for major psychiatric or neurological illness
* Major or unstable medical illness that might impact safety of the subject in the study
* Cannabis naive
* IQ less than 85
* Less than a high school diploma or its educational equivalent
* Pregnancy or lactation
* Major current or recent (<6 weeks) psychosocial stressors.

Inclusion Criteria FHN :

* Exposure to cannabis at least once in their lifetime
* Medically and psychiatrically healthy based on screening

Exclusion Criteria FHN:

* Having a family member with psychosis
* Current or lifetime major DSM-IV Axis I disorder
* Current or lifetime treatment (at least 6 months) with psychotropic medications for major psychiatric or neurological illness
* Major or unstable medical illness that might impact safety of the subject in the study
* Cannabis naive
* IQ less than 85
* Less than a high school diploma or its educational equivalent
* Pregnancy or lactation
* Major current or recent (<6 weeks) psychosocial stressors.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2014-01; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale for Schizophrenia (PANSS) | -30 min from administration of THC
  Positive, negative and general symptoms will be assessed using the positive, negative and general symptoms subscales of the PANSS.
Positive and Negative Symptom Scale for Schizophrenia (PANSS) | +80 min from administration of THC
  Positive, negative and general symptoms will be assessed using the positive, negative and general symptoms subscales of the PANSS.
Positive and Negative Symptom Scale for Schizophrenia (PANSS) | +150 min of administration of THC
  Positive, negative and general symptoms will be assessed using the positive, negative and general symptoms subscales of the PANSS.
Positive and Negative Symptom Scale for Schizophrenia (PANSS) | +240 min of administration of THC
  Positive, negative and general symptoms will be assessed using the positive, negative and general symptoms subscales of the PANSS.

SECONDARY OUTCOMES:
Clinician Administered Dissociative Symptoms Scale (CADSS) | -30 min, +15 min, +80 min, +150 min, +240 min
  Perceptual alterations will be measured using the CADSS. This is a scale consisting of 19 self-report items and 8 clinician-rated items (0=not at all, 4=extremely). The scale captures alterations in environmental/time/body perception, feelings of unreality, and memory impairment.
Visual Analog Scale (VAS) | -30 min, +15 min, +80 min, +150 min, +240 min
  Feeling states associated with cannabis intoxication will be measured using a self-reported visual analogue scale of four feeling states ("high", "anxious", "calm and relaxed", and "tired") associated with cannabis effects. Subjects will be asked to score the perceived intensity of these feeling states at that moment on a 11 mm line (0=not at all, 100=extremely). These data will be captured to validate that the experiment is relevant to cannabis effects.
Hopkins Verbal Learning Test (HVLT) | +50 min
  The HVLT is a 12 word list that is semantically organized. The task consists of 5 trials, an interference list, and free delayed recall and recognition. A different version of the AVLT will be administered on each test day and counterbalanced across subjects.
Psychotomimetic States Inventory (PSI) | -30 min, +240 min
  The PSI is a measure of drug induced psychotomimetic states. This self-report scale consists of 28 items rated 0 (not at all) to 3 (extremely) and will facilitate the characterization of a wide range of dissociative/hallucinatory phenomena as well as cognitive disorganization associated with the administration of THC.

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States